CLINICAL TRIAL: NCT07155512
Title: The Impact of a Bespoke Mindfulness Intervention for Registered Dietitians on Resilience, Burnout and Stress - A Cluster Randomised Control Trial
Brief Title: Impact of a Bespoke Mindfulness Intervention for Registered Dietitians on Resilience, Burnout and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMHS 70-1123
Record Dates: First submitted 2025-08-12; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Resilience, Psychological; Burnout, Professional; Stress, Psychological
Keywords: Registered Dietitian; Mindfulness; Randomised control trial; Resilience; Burnout; Stress; Mindfulness based intervention; Health personnel; Continuing professional development; Occupational health
MeSH Terms: conditions — Burnout, Professional; Stress, Psychological; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness based intervention (Experimental): Mindfulness based intervention (delivered synchronous online)
  Interventions: Behavioral: Mindfulness based intervention
- Waitlist control group (No Intervention): No intervention provided during the data collection period. Mindfulness based intervention delivered after data collection period.

INTERVENTIONS:
Behavioral: Mindfulness based intervention — A mindfulness intervention was designed especially for this study and delivered by a RD also qualified as a mindfulness teacher. The intervention was delivered synchronously online and consisted of 4 x 50 minute sessions delivered across 4 weeks.
  Arms: Mindfulness based intervention

SUMMARY:
The goal of this randomised control trial is to find out whether a mindfulness based intervention can improve mental well-being for Registered Dietitians (RD) in the UK. The main question it aims to answer is:

Can a mindfulness based intervention improve resilience amongst UK RDs?

Can a mindfulness based intervention reduce stress and burnout amongst UK RDs?

Researchers will compare participants who attend a structured mindfulness based intervention with a waitlist control group to see if there is a difference in outcome measures between the groups before the intervention, immediately after, 3 months after and 6 months after.

Participants in the intervention group will be invited to an online mindfulness course that was written especially for this study. Participants in both groups will be asked to complete surveys before the intervention, immediately after, 3 months after and 6 months after. Participants in the intervention group will also be invited to participate in a one to one interview to discuss their experiences, barriers and facilitators to mindfulness in dietetic practice.

ELIGIBILITY:
Inclusion Criteria:

* A Registered Dietitian currently practicing in the UK
* Willing and able to participate in 4 x 50 minute CPD sessions relating to mindfulness in dietetic practice (one session per week)
* Willing and able to complete all of the surveys (pre-intervention, immediately post, 3 months post and 6 months post intervention)

Exclusion Criteria:

* A diagnosis of a psychotic condition
* A diagnosis of epilepsy or asthma that is not well controlled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Resilience | Baseline, immediately after intervention (at the end of the last session of the 4 week intervention), 3 months post intervention, 6 months post intervention
  Measured using validated tool: Brief Resilience Scale. Scores range from 1-5. Higher scores = higher level of resilience. 1.00-2.99= Low resilience; 3.00-4.30 = Normal resilience; 4.31-5.00= High resilience.

SECONDARY OUTCOMES:
Burnout | Baseline, immediately post (this survey is administered at the end of the 4th and final session of the intervention, which was week 4), 3 months post, 6 months post intervention
  Measured using validated tool: Maslach Burnout Inventory, which has 3 domains which have the following scoring:
  Emotional Exhaustion (EE): </=17 low/more favourable; 18-29 moderate; >/= 30 high / least favourable Depersonalisation (DP): </=5 low/ more favourable; 6-11moderate; >/=12 high / least favourable Personal Accomplishment (PA): </=33 low / least favourable; 34-39moderate; </=40 high / most favourable
Stress | Baseline, immediately post intervention (this survey was given at the end of the 4th and final session of the intervention), 3 months post intervention, 6 months post intervention
  Measured using validated tool: Perceived Stress Scale - scores range from 0-40 with higher scores indicating higher levels of perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data collected in respect of 3 outcomes measured (resilience, burnout and stress) can be shared if required.

DOCUMENTS (1):
  • Informed Consent Form (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT07155512/ICF_000.pdf